CLINICAL TRIAL: NCT00832182
Title: An Open-labelled, Non-randomized, Multi-centre, Multinational Extension Trial Assessing the Safety of Insulin Aspart in Patients With Type I Diabetes Treated With a Basal-bolus Regimen
Brief Title: Examining the Long-term Safety of Insulin Aspart When Used as a Part of the Treatment for Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1229
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin aspart and neutral protamine Hagedorn insulin (Experimental)
  Interventions: Drug: insulin aspart; Drug: insulin NPH

INTERVENTIONS:
Drug: insulin aspart — Insulin aspart at breakfast, lunch and dinner time. Neutral protamine Hagedorn insulin at breakfast, lunch, dinner and bedtime. Injections were optional but at least one injection per day
Drug: insulin NPH — Insulin aspart at breakfast, lunch and dinner time. Neutral protamine Hagedorn insulin at breakfast, lunch, dinner and bedtime. Injections were optional but at least one injection per day

SUMMARY:
This trial is conducted in Europe and Asia. The aim of this clinical trial is to investigate the long-term safety of insulin aspart in the management of type 1 diabetes. An extension to the ANA/DCD/065 trial

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* The subject must have completed the ANA/DCD/065 trial

Exclusion Criteria:

* Impaired hepatic function
* Impaired renal function
* Total daily insulin requirements of more than 1.4 U/kg
* Cardiac problems
* Uncontrolled hypertension
* Known or suspected allergy to trial product or related products
* Current hypoglycaemic unawareness as judged by the investigator
* Known or suspect abuse of alcohol or narcotics
* Women breastfeeding or having the intention of becoming pregnant, or if judged not to be using adequate contraceptive measures (adequate measures are intrauterine device (IUD), oral contraception and barrier methods)
* Any condition that the Investigator and/or Sponsor feels would interfere with trial participation or evaluation of results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1999-12-22 (Actual); Primary Completion 2002-11-25 (Actual); Study Completion 2002-11-25 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic episodes and adverse events | at 3 and 6 months and at the end of the trial

SECONDARY OUTCOMES:
HbA1c | at 3 and 6 months and at the end of the trial
9-point blood glucose profile | at 3 and 6 months and at the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Ljubljana, Slovenia

REFERENCES:
- [Result] Cada DJ, Levien T, Baker DE. Insulin aspart. Hospital Pharmacy 2000; 35: 1221-1229
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com